CLINICAL TRIAL: NCT03160508
Title: A Prospective Study to Investigate Postoperative Real Life Weight Bearing Measured in Patients Treated With a Trochanter Fixation Nail Advanced (TFNA)
Brief Title: Trochanter Fixation Nail Advanced (TFNA) Weight Bearing
Status: Terminated | Type: Observational
Why Stopped: PCI decision due to technical issues
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: TFNA weight bearing
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2020-09

CONDITIONS: Femur Fracture
MeSH Terms: conditions — Femoral Fractures | interventions — Fracture Fixation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Fracture fixation with the TFNA — Fracture fixation with the TFNA

SUMMARY:
This study documents real life weight bearing in patients treated with a TFNA, who are allowed for immediate weight bearing as tolerated.

DETAILED DESCRIPTION:
Prospective data will be collected from 30 patients presenting a per- or inter-trochanteric fracture of the femur treated with the TFNA. Post-operatively patients will be asked to wear a sensor insole in their shoes for up to 3 months after surgical treatment. The sensor insole will be used in both feet and will not have any impact in patient's activities of daily living while allowing real time measurements of weight bearing.

In addition to weight bearing measurements, perceived pain (numeric rating scale), mobility (Parker Mobility Score and Time Up and Go Test) will be assessed at 6 and 12 weeks after surgical treatment and in conjunction with the standard (routine) of care follow up schedule. In order to investigate the relationship between these variables and the weight bearing measurements, patients or their care takers or assisting family members will be asked to document the daily use of the insole in a diary.

Finally, over the course of the study, anticipated adverse events (AE) that may affect the healing process will be collected. Special attention will be given to implant- or bone-related AEs. Images from patients with implant- or bone related AEs will be collected as per standard of care

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Patients treated with the TFNA; i.e. according to the technique guide and the indications for use, patients who presented any of the following conditions:

  * Stable or unstable pertrochanteric fractures
  * Intertrochanteric fractures
  * Basal neck fractures
  * Combinations of pertrochanteric, intertrochanteric, and basal neck fractures
* Patients who were able to walk before the fracture and are prescribed full weight bearing as tolerated post-surgery
* Ability to understand the content of the patient information / informed consent form
* Willingness and ability to participate in the study according to the clinical investigation plan
* Signed and dated ethical committee approved written informed consent according to the local regulations

Exclusion Criteria:

* Patients who are not allowed to full weight bearing as tolerated post-surgery
* Any condition, which impairs weight bearing (e.g. additional acute fracture on the ipsilateral and/or contralateral side, pain)
* Patients, who due to their condition, are in opinion of the Prinicipal Investigator (PI) unable to complete a reliable assessment
* Pregnancy or women planning to conceive within the study period
* Participation in any other medical device or medicinal product registry within the previous month that could, in opinion of the PI, influence the results of the present study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient matching all of the inclusion and none of the exclusion criteria at the respective study sites are invited to join the study.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Weight bearing | 3 months
  Time course of the weight bearing difference between the operated and the healthy legs within 3 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blauth, Prof., Principal Investigator — Medical University Innsbruck
Locations (2):
- Medical University Innsbruck, Innsbruck, Austria
- Kantonsspital Baselland, Binningen, Switzerland

IPD SHARING:
Plan to Share IPD: No